CLINICAL TRIAL: NCT01052909
Title: Randomized, 2-way Crossover, Bioequivalence Study of Glimepiride 1 mg Tablets and Amaryl 1 mg Tablets in Healthy Subjects Under Fasting Condition
Brief Title: Bioequivalence Study of Dr.Reddy's Laboratories Limited, Glimepiride Tablets 1 mg Under Fasting Condition
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Vice President - Research & Development, Dr. Reddy's Laboratories Limited
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 30286
Record Dates: First submitted 2010-01-19; First posted 2010-01-21 (Estimated); Last update posted 2010-01-21 (Estimated); Status verified 2010-01

CONDITIONS: Healthy
Keywords: Bioequivalence, Glimepiride, Crossover
MeSH Terms: interventions — glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Glimepiride (Experimental): Glimepiride tablets 1 mg of Dr. Reddy's Laboratories Limited
  Interventions: Drug: Glimepiride
- Amaryl (Active Comparator): Amaryl 1 mg tablets of Aventis Pharmaceuticals Inc
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Glimepiride — Glimepiride tablets 1 mg
  Other Names: Amaryl

SUMMARY:
The purpose of this bioequivalence study is to compare a test Glimepiride 1 mg tablets of Dr.Reddy's Laboratories Limited versus reference Amaryl 1 mg tablets of Aventis Pharmaceuticals Inc in healthy subjects, under fasting condition.

DETAILED DESCRIPTION:
The study was Single centre, randomized, single-dose, open-label,2-way crossover, bioequivalence study to compare a test Glimepiride 1 mg tablets of Dr.Reddy's Laboratories Limited versus Amaryl 1 mg tablets of Aventis Pharmaceuticals Inc in healthy subjects, under fasting condition.

ELIGIBILITY:
Inclusion Criteria:

* Male or non-child-bearing potential female,smoker and or non-smoker,18 years of age and older.
* Capable of consent.
* Non-child-bearing potential female subject:
* Post-menopausal state:absence of menses for 12 months prior to drug. administration or hysterectomy with bilateral oophorectomy at least 6 months prior to drug administration.
* Surgically sterile: hysterectomy, bilateral oophorectomy, or tubal ligation at least 6 months prior to drug administration.

Exclusion Criteria:

Subjects to whom any of the following applies will be excluded from the study:

* Clinically significant illnesses & surgery within 4 weeks prior to the administration of the study medication.
* Any clinically significant abnormality found during medical screening.
* Any reason which,in the opinion of the Medical Sub-Investigator,would prevent the subject from participating in the study.
* Abnormal laboratory tests judged clinically significant.
* Positive testing for hepatitis B and C or HIV at screening.
* ECG abnormalities (clinically significant) or vital sign abnormalities (systolic blood pressure lower than 90 or over 140 mmHg, diastolic blood pressure lower than 50 or over 90 mmHg, or heart rate less than 50 or over 100 bpm) at screening.
* BMI≥30.0.
* History of significant alcohol abuse within six months prior to the screening visit or any indication of the regular use of more than fourteen units of alcohol per week (l Unit=150 mL of wine, 360 mL of beer, or 45 mL of 40% alcohol).
* History of drug abuse or use of illegal drugs: use of soft drugs (such as marijuana) within 3 months prior to the screening visit or hard drugs (such as cocaine, phencyclidine [PCP] and crack) within 1 year prior to the screening visit or positive urine drug screen at screening.
* History of allergic reactions to glimepiride or other sulfonylureas (e.g. chlopropamide,gliclazide, tolbutamide and glyburide).
* History of allergic reactions to heparin.
* Use of any drugs known to induce or inhibit hepatic drug metabolism (examples of inducers: barbiturates, carbamazepine, phenytoin, glucocorticoids, rifampinlrifabutin; examples of inhibitors: antidepressants, cimetidine. diltiazem, erythromycin, ketoconazole, MAO inhibitors, neuroleptics, verapamil, quinidine) within 30 days prior to administration of the study medication.
* Use of an investigational drug or participation in an investigational study within 30 days prior to administration of the study medication. .
* Clinically significant history or presence of any clinically significant gastrointestinal pathology (e.g. chronic diarrhea. inflammatory bowel diseases), unresolved gastrointestinal symptoms (e.g. diarrhea, vomiting), liver or kidney disease, or other conditions known to interfere with the absorption, distribution, metabolism. or excretion of the drug.
* Any clinically significant history or presence of clinically significant neurological,endocrinal, cardiovascular, pulmonary, hematologic, immunologic, psychiatric, or metabolic disease.
* Use of prescription medication (including hormone therapy) within 14 days prior to administration of study medication or over-the-counter products (including natural food supplements, vitamins, garlic as a supplement) within 7 days prior to administration of study medication, except for topical products without systemic absorption.
* Difficulty to swallow study medication.
* Smoking more than 25 cigarettes per day.
* Any food allergy, intolerance, restriction or special diet that could, in the opinion of the Medical Sub-Investigator. contraindicate the subject's participation in this study.
* A depot injection or an implant of any drug within 3 months prior to administration of study medication.
* Donation of plasma (500 mL) within 7 days prior to drug administration. Donation or loss of whole blood prior to administration of the study medication as follows:
* 50 mL to 300 mL of whole blood within 30 days,
* 301 mL to 500 mL of whole blood within 45 days, or
* more than 500 mL of whole blood within 56 days prior to drug administration.
* Subjects with diabetes (including diabetes mellitus).
* Subjects with known serious hepatic impairments.
* Subjects with clinically significant presence or history of hypoglycemia.

Additional exclusion criteria for females only:

* Breast-feeding subject.
* Positive urine pregnancy test at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2003-12; Primary Completion 2003-12 (Actual); Study Completion 2003-12 (Actual)

PRIMARY OUTCOMES:
Bioequivalence study of Dr. Reddy's Laboratories Limited, Glimepiride tablets 1 mg under Fasting condition | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Girard, MD, Principal Investigator — Anapharm
Locations (1):
- Anapharm Inc, Sainte-Foy, Quebec, Canada